CLINICAL TRIAL: NCT02019628
Title: Enhancement of Natural Killer Cell Activity in Healthy Adults by Rice Bran Arabinoxylan Compound, a Novel Oligosaccharide
Brief Title: Enhanced Natural Killer Cell Activity and RBAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20090384
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Family Member
Keywords: NK cells cytotoxicity, dietary supplementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BRM4 at a dosage level of 1 gram/day (Experimental): 60-day trial of Rice Bran Arabinoxylan Compound (RBAC) at a dosage level of 1 gram/day.
  Interventions: Dietary Supplement: Rice Bran Arabinoxylan Compound (RBAC)
- BRM4 at a dosage level of 3 grams/day (Experimental): 60-day trial of Rice Bran Arabinoxylan Compound (RBAC) at a dosage level of 3 grams/day.
  Interventions: Dietary Supplement: Rice Bran Arabinoxylan Compound (RBAC)

INTERVENTIONS:
Dietary Supplement: Rice Bran Arabinoxylan Compound (RBAC) — Participants enrolled in the study will receive BRM4 at a dosage level of either 1 gram/day or 3 gram/day for the 60-day period. Subjects will be instructed to not consume any known immune-active pharmaceutical agents, nutritional supplements containing vitamins C and D, and/or any mushroom products for two weeks prior to having the baseline assessments and until the conclusion of the 60-day period. According to the company's literature, RBAC is a water soluble extract of rice bran that has been acted upon by an enzyme complex extracted from Shiitake mushroom. BRM4 contains: microcrystalline cellulose, hypromellose, sucrose fatty acid ester, gellan gum, and potassium acetate.

SUMMARY:
The present study investigated the effect of RBAC on natural killer cell activity (NKCA) and the production of cytokines and growth factors over 4 weeks among healthy adults.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the outcomes of a 60-day trial of Rice Bran Arabinoxylan Compound (RBAC) among adults. Specifically, subjects will participate in a two-group, randomized intervention that is based on a nutritional supplement made from a water soluble extract of rice bran that has been partially hydrolyzed by the action of a natural enzyme complex extracted from Shitake mushroom. One group will take 1 gram/day and the other group will take 3 gram/day to compare differences in outcomes between the two groups. We hypothesize that the 3 gram/day condition will demonstrate faster increases in outcomes compared to the 1 gram/day condition. The primary outcomes for this study will be Natural Killer (NK) cell activity, cytokines, total bilirubin, creatinine, and liver function tests. These outcomes will be compared between those subjects enrolled in the two treatment groups before and after 60 days.

No substantial psychological, medical, or social risks exist to the participants, other than minor discomfort associated with the venipuncture. Although all measures to protect confidentiality will be put in place, the possibility exists that electronic data could be jeopardized. In the remote case that such event occurs, it will be immediately reported to the IRB.

The components of RBAC should be harmless without significant food allergies. No serious, untoward side effects have been reported to the company by consumers nor observed during previous human studies. If any side effect does occur, the remedy is to discontinue until asymptomatic, and then reintroduce at 1/4 dosage, increasing by the same amount every 2 days, if uneventful, until full dosage is achieved. Dr. Ali will provide additional follow-up and consultation with any subject who experiences an untoward side effect.

A toxicology search for each component reveals no unique toxicity characteristic of the materials. As reported by Daiwa Health Development, the manufacturer of the product, thousands of people currently use RBAC (under the trade names BRM4 and PeakImmune 4), and Daiwa is unaware of significant toxicities. Daiwa applies the latest scientific methods to ensure the value and safety of their raw materials. Daiwa products are manufactured in state-of-the-art facilities, under strict quality control and environmental protection standards.

Participants will incur no additional appreciable psychological or social risks by participating in this study, although they may undergo psychological and physical discomfort sometimes. The process of interviewing during the assessment may cause discomfort. Discomfort or fatigue may also be experienced in completing the assessment battery.

Alternatives to this study for enhancing immune system functioning include prescription medications, exercise, dietary modification, and other nutritional supplements. The risks of medications can be very significant, including life-threatening, but the risk of taking nutritional supplements is not totally understood, since they are not regulated by the US Food and Drug Administration. Medications and nutritional supplements, as part of a change in lifestyle behaviors, may also prove to be beneficial for immune system functioning, but their long-term use has unknown consequences.

The information obtained in this study will help in determining the efficacy of using a rice bran extract nutritional supplement for enhancing immune system outcomes. By participating in the study, subjects may experience improved NK cell activity and cytokine functioning. The risk of participating in this study is reasonable because of the potential enhancements in immune system functioning with improved nutritional status.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men ages 18 years and over.
2. Interest in participating in a novel nutritional supplement program.
3. Willingness to follow recommendations.

Exclusion Criteria:

1. Currently enrolled in another research trial for investigative nutritional or other therapies thought to have an impact on immune system functioning.
2. Unable to consent to the study.
3. Women who are pregnant or are attempting conception, especially in the presence of a history of recurrent spontaneous abortion.
4. Other medical complications that might preclude one from participating in the study, i.e., recent heart attack or stroke or chronic kidney disease.
5. Currently taking immunomodulatory medication, i.e. interferon.
6. Currently taking other medications thought to have an impact on immune system functioning, i.e., chemotherapeutic agents.
7. Known allergy to rice, rice bran, or related food products.
8. Known allergy to mushrooms or related food products.
9. History of malignancies related to the NK cell line, including: NK cell leukemias and T-cell large granular lymphocyte leukemias, NK-cell lymphoproliferative disease of granular lymphocytes, and NK cell lymphomas, e.g., nasal and nasal-like NK/T-cell lymphomas.
10. Current smoker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Immune Functioning - NK Cell activity | 60 days
  NK Cell activity at baseline, 48 hours, 1 week, 1 month, and 2 months.
Immune Functioning - Cytokines | 60 days
  Cytokines at baseline, 1 month, and 2 months.

SECONDARY OUTCOMES:
Bilirubin | 60 days
  Bilirubin at baseline, 48 hours, 1 week, 1 month, and 2 months.
Blood Pressure and Heart Rate | 60 days
  Blood pressure and heart rate at baseline and 2 months.
Physical Activity | 60 days
  Physical activity will be assessed at baseline and 2-months follow-up by the Stanford 7-day Activity Recall. This instrument assesses the amount (number of hours) of moderate, physically challenging, and very physically challenging activities over the past 7 days. This instrument provides useful estimates of habitual physical activity for research, significantly agrees with daily self-report of physical activity, and has been validated for use in community settings.
Functional Health and Well-being | 60 days
  The SF-36v2™ Health Survey provides psychometrically-based physical and mental health summary measures and a preference-based health utility index. It is a generic measure that does not target a specific age, disease, or treatment group and will be assessed at baseline and 2-months follow-up.
Creatinine | 60 days
  Creatinine at baseline, 48 hours, 1 week, 1 month, and 2 months.
Liver Function Tests | 60 days
  Liver Function Tests at baseline, 48 hours, 1 week, 1 month, and 2 months.
Body Mass Index | 60 days
  Body weight and height to calculate body mass index (BMI) at baseline and 2 months.
Percent Body Fat | 60 days
  Skinfold caliper assessment to calculate percent body fat at baseline and 2 months.
Waist to Hip Ratio | 60 days
  Waist and hip circumference to calculate waist to hip ratio at baseline and 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: John E. Lewis, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami CRB, Miami, Florida, United States